CLINICAL TRIAL: NCT06194903
Title: Randomized Experimental Pilot Study Evaluating Isopropyl Alcohol and UVC Rays in Disinfection of Cell Phones of Healthcare Workers.
Brief Title: Randomized Pilot Study Evaluating Isopropyl Alcohol and UVC Rays in Disinfection of Cell Phones
Acronym: SaniPhone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6015
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Cross Infection
Keywords: cross infection; high touch surfaces; cellphone; disinfection; isopropyl alcohol; UVC
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cellphones treated with isopropyl alcohol wipes (Experimental)
  Interventions: Device: isopropyl alcohol wipes
- Cellphones treated with UVC box (Experimental)
  Interventions: Device: UVC box

INTERVENTIONS:
Device: isopropyl alcohol wipes — cellphones will be sanitised with isopropyl alcohol wipes and total bacterial load will be assessed immediately before sanitation, immediately after sanitation and 3 hours after sanitation.
  Arms: Cellphones treated with isopropyl alcohol wipes
Device: UVC box — cellphones will be sanitised in a UVC box and total bacterial load will be assessed immediately before sanitation, immediately after sanitation and 3 hours after sanitation.
  Arms: Cellphones treated with UVC box

SUMMARY:
Cell phones have become a fundamental accessory of our lives and clinical practice, often kept in contact with the body. Since most modern smartphones are equipped with touch screens, they can serve the function of reservoirs for pathogenic microorganisms; moreover, they can be the means of transmission of such microorganisms from the environment to humans.

A number of observational studies are available in the literature evaluating the effectiveness of various sanitization methods in reducing the bacterial load of high-touch devices, both chemical and physical.

To our knowledge, no real-world evidence is available comparing the residual effect of the two methods on the bacterial load of cell phones, since all available studies are carried out in the laboratory, with inoculums of predetermined bacterial loads whose suppression by the disinfectant is monitored over time, and involve laptops, tablets and keyboards.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthcare provider in the departments of Neonatology, Geriatric Internal Medicine, Nephrology, Anesthesia, Resuscitation, Intensive Care Unit at Fondazione Policlinico Universitario "A.Gemelli" IRCCS
* Own a smartphone
* Carry one's smartphone for the duration of the work shift (8 hours)
* Give consent to participate in the study
* Be willing to report 3 hours after sanitisation for follow-up sampling

Exclusion Criteria:

* Not to be a healthcare worker in the departments of Neonatology, Geriatric Internal Medicine, Nephrology, Anesthesia, Resuscitation, Intensive Care Unit at Fondazione Policlinico Universitario "A.Gemelli" IRCCS
* Not to be on work shift during surveys
* Not to carry one's smartphone for the duration of the work shift (8 hours)
* Not to give consent to participate in the study
* Not to be willing to report 3 hours after sanitisation for follow-up sampling

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Average total bacterial load at 3 hours after sanitization | Samples will be collected immediately before and immediately after sanitisation and 3 hours after sanitisation.
  The primary objective of the pilot study is to obtain preliminary data on the average total bacterial load at 3 hours after the sanitization intervention (70% isopropyl alcohol wipes or UVC box). These data will allow appropriate sizing of a subsequent trial to evaluate whether, on the cell phones of health care workers at the Fondazione Policlinico Universitario "A. Gemelli" IRCCS, wipes impregnated with 70% isopropyl alcohol are more effective than UVC ray boxes in reducing total bacterial load at 3 hours after sanitization for both isopropyl alcohol wipes and UVC box

SECONDARY OUTCOMES:
Change in the average total bacterial load at 3 hours after sanitization | Samples will be collected immediately before and immediately after sanitisation and 3 hours after sanitisation
  Explore the change in the average total bacterial load at 3 hours after sanitization interventions compared with the value recorded before sanitisation for both isopropyl alcohol wipes and UVC box.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A. Gemelli" IRCCS, Rome, Italy